CLINICAL TRIAL: NCT03424655
Title: Use of Intracanal Cryotherapy on Post-endodontic Pain After Single-visit RCT Using Manual and Reciprocating Systems When Apical Patency is Conserved.
Brief Title: Post-endodontic Pain After Single-visit Root Canal Treatment
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Paredes Vieyra (Other)
Responsible Party: Sponsor-Investigator, Jorge Paredes Vieyra, Dr. Jorge Paredes Vieyra D.D.S., MsC, PhD, Universidad Autonoma de Baja California
Organization: Universidad Autonoma de Baja California (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: endodontic pain 2018
Record Dates: First submitted 2018-01-18; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Relate Post-endodontic Pain
Keywords: post -endodontic pain; endodontic pain; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: teeth selected for conventional RCT for prosthetic reasons detected with only vital pulps. Of the sample of 224 teeth, 56 were selected to the 4 instrumentation methods. For hand instrumentation, Balanced Force were used. All canals were clean and shaped with hand Flex-R files (fMoyco/Union Broach, York PA, USA). For mechanical shaping, all instruments were used with a micro motor (VDW, Munich Germany). Twisted files adaptive, WaveOne and Reciproc instruments. Final irrigation with cold (6oC) 17% EDTA served as a lubricant.
Who Masked: Participant, Investigator
Masking Description: Certified endodontists trained in the procedures, devices, and systems investigated took part in the research. All experts tracked a pre-established procedure for the Balanced Force technique, Twisted File Adaptive, WaveOne, and Reciproc instrument systems.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group TFA (Experimental): Twisted files were used serially with a single controlled motion according to the manufacturer's instructions.
  Interventions: Procedure: Twisted File Adaptive
- Group BF (Experimental): The root canals were cleaned and shaped using a #40 instrument for thin or curved canals and a #55 file for widespread canals.
  Interventions: Procedure: Balance Force
- Group WON (Experimental): WaveOne files was used to prepare narrow, straight and curved canals, and a file (40.08) was used for large and wide canals.
  Interventions: Procedure: WaveOne
- Group REC (Experimental): Reciproc instrument was used in thin and curved RC, and R40 files (40.06) were used in wide canals.
  Interventions: Procedure: Reciproc technique

INTERVENTIONS:
Procedure: Twisted File Adaptive — Twisted file adaptive SM1 (size 20, .04 taper) and SM2 (size 25, .06 taper) were used serially with a single controlled motion according to the manufacturer's instructions.
  Arms: Group TFA
Procedure: Balance Force — Flex-R files sizes 15-45 taper .02 were used according to the technique
  Arms: Group BF
Procedure: WaveOne — WaveOne instrument was used to prepare narrow, straight and curved canals, and file (40.08) was used for large canals.
  Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.
  Arms: Group WON
Procedure: Reciproc technique — Reciproc files were used in wide canals. Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.
  Arms: Group REC

SUMMARY:
The goal of this research was to relate the occurrence of post-endodontic pain after single-visit RCT using Balanced Force technique and three reciprocating system when AP is conserved. Methodology: All 224 patients had upper or lower molar, premolar or anterior teeth selected for conventional RCT for prosthetic reasons detected with only vital pulps. Of the sample of 224 teeth, 56 were selected to the 4 instrumentation methods. For hand instrumentation, Balanced Force were used. All canals were clean and shaped with hand Flex-R files (fMoyco/Union Broach, York PA, USA). For mechanical shaping, all instruments were used with a micro motor (VDW, Munich Germany). Twisted files adaptive, WaveOne and Reciproc instruments. Final irrigation with cold (6oC) 17% EDTA served as a lubricant.

DETAILED DESCRIPTION:
This clinical research took place at the University Autonomous of Baja California, School of Dentistry, Tijuana, Mexico. The subjects review committee accepted the research, and conducted in accordance with ethical principles (including the World Medical Association Declaration of Helsinki).

The principal inclusion parameters were absence of radiographic sign of apical periodontitis and a diagnosis of irreversible pulpitis (IP) established by affirmative response to hot and cold examinations.

Thermal pulp examination was achieved by the corresponding author, and radiographic analysis was established by 3 certified endodontists. Clinical requirements were established on the next conditions: 1) The purposes and necessities of the research were spontaneously accepted. 2) Clinical Management was pointed to patients in physical and mental well-being. 3) All teeth had vital pulps and absence of apical periodontitis. 4) Positive thermal stimulation with EndoIce (Hygenic Corp, Akron, OH). 5) Teeth with enough coronal structure for rubber dam isolation. 6) No RCT done before the research. 7) No painkillers or antibiotics used 7 days' prior the clinical events started.

Exclusion parameters were the necessity for retreatment, gravidity, impossibility to obtain patient's approval, patients who didn't complete inclusion necessities, a history of medication for chronic pain or those compromising the immune response, patients younger than 18 years and the existence of mishaps or difficulties during RCT (calcified canals, impracticality of achieving AP in any canal).

Patient selection Two hundred and twenty four of 245 patients (126 women and 98 men) aged 18-65 years were incorporated in this research (Fig. 1). Sample size estimate was achieved according with a method for this specific purpose (Cochran's method, 1986). Therefore, the 56 teeth allocated to each group were adequate to confirm an essential sample.

Random Selection of instrumentation groups. Of the sample of 224 teeth, 56 were selected to the 4 instrumentation methods. The study strategy included 3 experts; each expert prepared 56 teeth, 14 per technique.

Treatment Protocol The standard method involved the following steps: Access was gotten; REDTA (Roth International, Chicago, IL) lubricant was located at the entry of the canals. Determination of WL was first determined with a #15 k-file and the Root ZX electronic device (J Morita, Irvine CA, USA), following by subtracting 0.5 mm from the measurement, which was calculated with the assistance of a metallic ruler. With digital radiographic confirmation (Schick Technologies, NY, USA). A glide path to the WL was then established.

For hand instrumentation, Balanced Force were used. All canals were clean and shaped with hand Flex-R files (fMoyco/Union Broach, York PA, USA). Gates-Glidden burs (Dentsply Maillefer) sizes #2 and #3 were used at the entry of the canals. For mechanical shaping, all instruments were used with a micro motor (VDW Silver Reciproc Motor). Torque and rotation were established independently for each instrument method used. Twisted file adaptive, WaveOne and Reciproc instruments were used in continuous brushing rotary motion and reciprocating mode respectively.

Group TFA. SM1 (size 20, .04 taper) and SM2 (size 25, .06 taper) files were used serially with a single controlled motion according to the manufacturer's instructions.

Group BF. For the Balanced force group, the root canals were cleaned and shaped using a #40 instrument for thin or curved canals and a #55 file for widespread canals.

Group WON. For the WaveOne group, a file (25.08) was used to prepare narrow, straight and curved canals, and a file (40.08) was used for large and wide canals.

Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.

Group REC. R25 (25.08) instrument was used in thin and curved RC, and R40 files (40.06) were used in wide canals. Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.

Hand and rotary files were employed in just 1 tooth (single use) and then excluded. AP was conserved through all the procedures used by using a #10 K-type file at WL.

After instrumentation phase, pulp chamber was rinsed with 1 mL 2.6% NaOCl, agitated ultrasonically. Ultrasonic activation was performed using an Irrisafe ultrasonic 20.00 tip (Satelec, M erignac, France) at 50% power of the MiniEndo ultrasonic unit (Kerr Endo) to place the tip 3 mm from the WL for 30 seconds per canal. Then, each experimental group received a final irrigation with cold (6oC) 17% EDTA gently delivered to the WL using a cold (6oC) sterile metallic micro cannula attached to the Endovac negative pressure irrigation system (Kerr Endo) for three minutes to eliminate the smear layer and reduce post-endodontic pain. Caution was taken to ensure that the micro cannula would suction correctly by detecting the system's transparent evacuation tube. In case there was any obstruction, the micro cannula was instantly substituted.

Repeat of WL was established again by using EAL as describe before using #35, #40 and # 45 files.

The root canals were then desiccated with disinfected paper cones and filled at the same visit. Gutta-percha cones (Dentsply Maillefer) were laterally compacted with #20 nickel-titanium spreaders (Dentsply Maillefer) and AH-plus sealer (Dentsply Maillefer). Entrance openings of anterior teeth were etched and repaired with Fuji IX (GC Corp, Tokyo, Japan). For posterior teeth, a rebuilding was placed with the same method.

Assessment of Post-endodontic pain and Statistical Analysis Patients were informed of the probable incidence of pain for days following RCT and received a survey form to be finished and returned three days after. In it, they proof the occurrence or nonappearance of post-endodontic pain, its period and level of distress rated as follows: mild pain: any discomfort of any duration that does not require treatment; moderate pain: pain that requires and is relieved with analgesics; and severe pain: any pain that is not calmed with treatment (analgesics).

Outcomes were examined with the Chi-Square for the occurrence of post-endodontic pain, and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* The principal inclusion parameters were absence of radiographic sign of apical periodontitis and a diagnosis of irreversible pulpitis (IP) established by affirmative response to hot and cold examinations.

Thermal pulp examination was achieved by the corresponding author, and radiographic analysis was established by 3 certified endodontists. Clinical requirements were established on the next conditions: 1) The purposes and necessities of the research were spontaneously accepted. 2) Clinical Management was pointed to patients in physical and mental well-being. 3) All teeth had vital pulps and absence of apical periodontitis. 4) Positive thermal stimulation with EndoIce (Hygenic Corp, Akron, OH). 5) Teeth with enough coronal structure for rubber dam isolation. 6) No RCT done before the research. 7) No painkillers or antibiotics used 7 days' prior the clinical events started.

Exclusion Criteria:

* Exclusion parameters were the necessity for retreatment, gravidity, impossibility to obtain patient's approval, patients who didn't complete inclusion necessities, a history of medication for chronic pain or those compromising the immune response, patients younger than 18 years and the existence of mishaps or difficulties during RCT (calcified canals, impracticality of achieving AP in any canal).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Use of intracanal cryotherapy on post-endodontic pain after single-visit RCT using manual and reciprocating systems when Apical Patency is conserved. | 24 hrs
  Relate the post-endodontic pain after single-visit After the root canal treatment with Balanced Force technique and three reciprocating system.

SECONDARY OUTCOMES:
Use of intracanal cryotherapy on post-endodontic pain after single-visit RCT | 24 hrs
  A final irrigation after root canal treatment was made with cold 3cc of (6oC) 17% EDTA gently delivered to the WL using a cold (6oC) sterile metallic micro cannula.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Clemente, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No
This clinical research took place at the University Autonomous of Baja California, School of Dentistry, Tijuana, Mexico. The subjects review committee accepted the research, and conducted in accordance with ethical principles (including the World Medical Association Declaration of Helsinki).

REFERENCES:
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729